CLINICAL TRIAL: NCT01526837
Title: A Dose-Escalating Phase I Study for Safety and Tolerability of Bevacizumab in Collagen Delivery Vehicle Administered Into the Tumor Resection Cavity in Subjects With Glioblastoma Multiforme at First Recurrence
Brief Title: Bevacizumab (Avastin) Into the Tumor Resection Cavity in Subjects With Glioblastoma Multiforme at First Recurrence
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Investigators decision
Sponsor: Brain & Spine Surgeons of New York (Other)
Responsible Party: Principal Investigator, John Abrahams, M.D., Associate Professor of Neurosurgery, Brain & Spine Surgeons of New York
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BSSNY-B-001
Record Dates: First submitted 2011-11-05; First posted 2012-02-06 (Estimated); Last update posted 2017-07-12 (Actual); Status verified 2017-07

CONDITIONS: Glioblastoma Multiforme
Keywords: Brain tumor; GBM; Brain cancer
MeSH Terms: conditions — Glioblastoma; Brain Neoplasms | interventions — Bevacizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- bevacizumab (Avastin) (Experimental): Open-label, dose-escalating study conducted in cohorts of 1-3 patients treated at increasing doses of bevacizumab in the dose range of 1-25mg/Ml. A maximum of 24 subjects will be treated in this study (up to 8 cohorts of 3 subjects).
  Interventions: Drug: Avastin

INTERVENTIONS:
Drug: Avastin — Topical Avastin plus Collagen Sponge placed in surgical cavity after resection of recurrent brain tumor. Dosing range: 0.25 mg/ml - 25 mg/ml.

SUMMARY:
This is a phase 1b study for safety and tolerability of bevacizumab(Avastin)administered into the tumor resection cavity in subjects with Glioblastoma Multiforme (GBM) at first recurrence.

ELIGIBILITY:
Inclusion Criteria:

1. Recurrent Glioblastoma
2. At least 12 weeks expected survival (KPS >60)
3. 18 years of age or older
4. Able and willing to participate

Exclusion Criteria:

1. Any prior diagnosis of any other cancer or other concurrent malignancy.
2. Planned use or current use of other investigation therapy.
3. Systemic autoimmune disease
4. HIV positive
5. Concurrent life threatening disease
6. Impaired organ function
7. Active infection
8. Inadequately controlled hypertension
9. Congestive heart failure
10. Myocardial infection/unstable angina within 6 months
11. Stroke within 6 months
12. Pheripheral vascular disease
13. History of abdominal fistula/gastrointestinal performation
14. Non-healing wound
15. Coagulation disease
16. Known allergy to study treatments
17. Pregnant or lactating

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2011-10; Primary Completion 2012-01 (Actual); Study Completion 2012-01 (Actual)

PRIMARY OUTCOMES:
Maximum Tolerated Dose of bevacizumab (Avastin) following local administration. | 4 weeks

SECONDARY OUTCOMES:
Number of Adverse Events | 12 months
  All adverse events will be recorded in the case report form.
Progression Free Survival | 12 months
  Patients will be followed for survival as well as disease progression for 12 months after treatment.

CONTACTS AND LOCATIONS:
Overall Officials: John Abrahams, MD, Principal Investigator — Brain & Spine Surgeons of New York; Jan Strack, Study Director — BSSNY
Locations (1):
- Brain & Spine Surgeons of New York, White Plains, New York, United States